CLINICAL TRIAL: NCT05966389
Title: Assessment of Cerebral Microcirculation, Blood-brain Barrier, and Cerebral Oxygenation Damage in Patients with Cardiac Arrest Using Functional MRI
Brief Title: Functional MRI to Assess Brain Damage in Cardiac Arrest Patients
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Tang Ziren, Professor, Capital Medical University
Other Study IDs: 2023-6-21-8
Record Dates: First submitted 2023-07-18; First posted 2023-07-28 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Arrest; Brain Injuries
Keywords: Cardiac arrest; functional Magnetic Resonance Imaging; cerebral microcirculation; blood-brain barrier; cerebral oxygenation
MeSH Terms: conditions — Heart Arrest; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
This is a single-center, observational study. Patients after successful cardiopulmonary resuscitation (CPR) will be transferred to the emergency intensive care unit for further standardized management. After successful return of spontaneous circulation (ROSC) for 72h and hemodynamics remained stable for 24h, the post-resuscitated patients underwent functional magnetic resonance imaging (fMRI) examination. During the examination, the supervising physician accompanied the patient and monitored the patient's vital signs using a magnetic resonance monitoring system (Siemens Healthcare Prism, Germany). Patients who are on ventilators are mechanically ventilated using a magnetic ventilator (HAMILTON-MRI, USA). In additional to conventional sequences, fMRI is performed for diffusion-prepared pseudo-continuous arterial spin labeling (DP-pCASL) and blood oxygenation level dependent functional magnetic resonance imaging (BOLD-fMRI). These MRI sequences allow quantitative assessment of the patients' cerebral microcirculation, blood-brain barrier, and cerebral oxygenation status. Patients will be followed up for neurologic prognosis according to the Modified Rankin Scale (mRS) at 6 months after disease onset.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years.
* sustained hemodynamic stability for ≥24h.
* the patients were unconscious and not able to obey verbal commands.
* Advanced life support and target temperature management within 6 hours of return of spontaneous circulation (ROSC).

Exclusion Criteria:

* Patients with hemodynamic instability.
* Patients who could not complete cranial MRI examination for special reasons.
* Patients during pregnancy.
* Patients who combined traumatic brain injury, stroke, cerebral hemorrhage and other diseases.
* Patients whose family members did not agree to be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after successful cardiopulmonary resuscitation (CPR) were transferred to the emergency intensive care unit for further standardized management.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Neurologic prognosis | 6 months
  Patients will be followed up for neurologic prognosis according to the Modified Rankin Scale (mRS) at 6 months after disease onset.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chaoyang hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: The de-identified survey data will be made available for research purposes by contacting the corresponding authors

REFERENCES:
- [Derived] Shao R, Wang T, Hang C, An L, Wang X, Zhang L, Yu J, Shan Z, Yang Q, Tang Z. Alteration in early resting-state functional MRI activity in comatose survivors of cardiac arrest: a prospective cohort study. Crit Care. 2024 Aug 2;28(1):260. doi: 10.1186/s13054-024-05045-4. PMID 39095884